CLINICAL TRIAL: NCT04524676
Title: Construction and Evaluation of the Early Identification and Individualized Treatment for Oxaliplatin-induced Portal Hypertension
Brief Title: Oxaliplatin-induced Portal Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLAEGV
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Gastroesophageal Varices Hemorrhage; Colorectal Cancer; Received Oxaliplatin-based Chemotherapy
Keywords: portal hypertension; gastroesophageal variceal bleeding; colorectal carcinoma; splenomegaly; oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms; Hypertension, Portal; Splenomegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized Treatment Group (Experimental)
  Interventions: Procedure: Individualized Treatment

INTERVENTIONS:
Procedure: Individualized Treatment — Patients under evaluation including hepatic venous pressure gradient (HVPG) and contrast-enhanced computed tomography of portal venous. For those patients with a HVPG ≥12mmHg or with extraluminal para-gastric vein will under transjugular intrahepatic portosystemic shunt and others receive endoscopic treatment.

SUMMARY:
Oxaliplatin has been used as the first choice for the adjuvant chemotherapy of colorectal cancer and it has significantly improved the outcomes in patients with colorectal cancer. However, hepatotoxicity is the potentially problematic adverse effect of oxaliplatin. The pathological evaluation of non-tumoral liver from patients with advanced colorectal cancer undergoing neoadjuvant oxaliplatin-based treatment has provided histological evidence of hepatic sinusoidal injury. Oxaliplatin-induced sinusoidal injury can persist for more than 1 year after the completion of chemotherapy, and the increase in splenic volume may be a predictor of irreversible sinusoidal damage. In this current study, we aim to evaluate the efficacy of individualized treatment in patients with oxaliplatin-induced gastroesophageal varices after colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent
* Male or female patients aged 18-75
* diagnosed as portal hypertension by contrast-enhanced computed tomography
* and confirmed gastroesophageal varices by upper digestive endoscopy;
* had a history of oxaliplatin-based chemotherapy after colorectal cancer surgery;

Exclusion Criteria:

* combined known etiologies of chronic liver disease, including hepatitis, primary biliary cirrhosis, schistosomiasis, and non-alcoholic fatty liver disease.
* with colorectal cancer required further anti-tumor treatment
* Other factors judged by the investigator that may affect the safety of the subject or the compliance of the trial. Such as serious illnesses (including mental illness) that require combined treatment, serious laboratory abnormalities, or other family or social factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-08-31 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
1-year rebleeding rate | 1 year
  1-year rebleeding rate

SECONDARY OUTCOMES:
1-year death rate | 1 year
  1-year death rate
Complications of portal hypertension | 1 year
  The occurrence of complications of portal hypertension including ascites, liver failure, et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology and Hepatology, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Huang X, Li F, Wang L, Xiao M, Ni L, Jiang S, Ji Y, Zhang C, Zhang W, Wang J, Chen S. Endoscopic treatment of gastroesophageal variceal bleeding after oxaliplatin-based chemotherapy in patients with colorectal cancer. Endoscopy. 2020 Sep;52(9):727-735. doi: 10.1055/a-1157-8611. Epub 2020 May 7. PMID 32380558
- [Result] Aloia T, Sebagh M, Plasse M, Karam V, Levi F, Giacchetti S, Azoulay D, Bismuth H, Castaing D, Adam R. Liver histology and surgical outcomes after preoperative chemotherapy with fluorouracil plus oxaliplatin in colorectal cancer liver metastases. J Clin Oncol. 2006 Nov 1;24(31):4983-90. doi: 10.1200/JCO.2006.05.8156. PMID 17075116
- [Result] Iwai T, Yamada T, Koizumi M, Shinji S, Yokoyama Y, Takahashi G, Takeda K, Hara K, Ohta K, Uchida E. Oxaliplatin-induced increase in splenic volume; irreversible change after adjuvant FOLFOX. J Surg Oncol. 2017 Dec;116(7):947-953. doi: 10.1002/jso.24756. Epub 2017 Sep 6. PMID 28876454
- [Result] Ward J, Guthrie JA, Sheridan MB, Boyes S, Smith JT, Wilson D, Wyatt JI, Treanor D, Robinson PJ. Sinusoidal obstructive syndrome diagnosed with superparamagnetic iron oxide-enhanced magnetic resonance imaging in patients with chemotherapy-treated colorectal liver metastases. J Clin Oncol. 2008 Sep 10;26(26):4304-10. doi: 10.1200/JCO.2008.16.1893. PMID 18779617